CLINICAL TRIAL: NCT06015295
Title: A Pilot Study to Assess the Clinical Utility of 18F-Fluciclovine (Axumin) PET-CT for Detecting True-versus Pseudo-Progression of Brain Metastases on Immunotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0159; NCI-2024-09643 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-Fluciclovine (Axumin) (Experimental): Participants are expected to be in this research study for about 6-12 months. Participants will have up to 6 visits for screening tests, Axumin PET-CT scans, and information collection.
  Interventions: Diagnostic Test: 18F-Fluciclovine (Axumin); Diagnostic Test: Pet Scan

INTERVENTIONS:
Diagnostic Test: 18F-Fluciclovine (Axumin) — Given by Injection
Diagnostic Test: Pet Scan — Scans

SUMMARY:
To learn if 18F-Fluciclovine (Axumin) PET-CT scans can be used to better detect brain metastatic lesions in patients who are receiving immunotherapy.

DETAILED DESCRIPTION:
Primary Objective:

* To assess the diagnosis accuracy of 18F-Fluciclovine (Axumin) PET-CT in detecting true- versus pseudo-progression of brain metastatic lesions in patients on immunotherapy.

Accuracy is defined as the number of concordant cases between Axumin PET-CT and the gold standard truth divided by the total sample size.

Secondary Objectives

* To assess diagnosis accuracy of Axumin PET-CT in detecting true- versus pseudo-progression of brain metastatic lesions in patients on immunotherapy by additional accuracy measures including sensitivity, specificity, negative predictive value and positive predictive value.
* To evaluate the added clinical usefulness of Axumin PET-CT for imaging patients with metastatic brain lesion(s).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of Axumin in pediatric patients, patients <18 years of age are excluded from this study.
2. ECOG performance status ≤2 (Karnofsky ≥60%,).
3. Willingness to participate in the study and ability to provide written informed consent.
4. Patients must have documented brain metastatic lesion(s) in the medical record.
5. On active immunotherapy for the diagnosed malignancy. Concurrent other treatment is allowed. Immunotherapy and other treatment regimens are determined by treating physicians as per standard clinical practice.
6. Patients with at least one metastatic brain lesion showing suspected pseudoprogression on SoC imaging modality (such as CT, or MRI, or FDG PET-CT, or DOTATATE PET/CT, or PSMA PET/CT).
7. The suspected pseudoprogresson can be determined by imaging physician (such as neuroradiologists and/or nuclear medicine physicians) and/or treating physicians (usually are oncologists). Ideally, the target/index lesion should be measurable (at discretion of investigator imaging physicians) and feasible for series follow up and comparison at imaging physician's discretion.
8. Ability and willingness to undergo another follow up Fluciclovine PET/CT, usually within 60 days of SoC follow up imaging modality.
9. Ability and willingness to undergo biopsy if needed per standard of care.
10. Estimated life expectancy of at least 3 months as determined by the investigator or treating physician.

Exclusion Criteria:

1. Pregnant or breastfeeding during participation in the study are excluded because: There is no information on the risk of adverse developmental outcomes in pregnant women or animals with the use of Fluciclovine F18. All radiopharmaceuticals, including Axumin, have the potential to cause fetal harm depending on the fetal stage of development and the magnitude of the radiation dose; There is no information on the presence of Fluciclovine F18 in human milk, the effect on the breastfed infant, or the effect on milk production.
2. History of severe allergic reactions to Axumin PET radiopharmaceuticals. Mild to moderate reactions that can be controlled by medications prior to the scheduled PET/CT are acceptable.
3. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
4. Unable to lie flat during or tolerate PET-CT
5. Contraindications to Axumin Injection have not been established in humans. None are known or have been observed in nonclinical or clinical studies performed to date.
6. Subjects with any medical condition or circumstance that the investigator believes may compromise the safety or compliance of the subject to produce reliable data or completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org